CLINICAL TRIAL: NCT03183466
Title: Prospective Randomized Clinical Trial of Arthroscopic Repair Versus Debridement for Subscapularis Tendon Tear More Than 1/2 to Entire 1st Facet (Representing 1/3 to More Than 1/3 Tear of Subscapularis Entire Footprint)
Brief Title: Do You Arthroscopic Repair for Subscapularis Tendon Tear, Which Accounts for More Than Half of the 1st Facet? Or do You Perform Debridement?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 2011-11-029-025
Record Dates: First submitted 2017-05-30; First posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-05

CONDITIONS: Subscapularis Tendon Tear; Arthroscopic Repair; Arthroscopic Debridement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients included in inclusion criteria (Experimental)
  Interventions: Procedure: arthroscopic repair; Procedure: arthroscopic debridement

INTERVENTIONS:
Procedure: arthroscopic repair
Procedure: arthroscopic debridement

SUMMARY:
The purpose of this study was to randomly classify the upper third of the subscapularis in 1/2 of the rupture patients as preoperative group (arthroscopic and arthroscopic debridement group) and the difference between clinical and clinical scores.

DETAILED DESCRIPTION:
The degree of rupture that is an adaptation of arthroscopic surgery is now known to be about one-third to one-half of a rupture. However, the most controversial case is the one-third to one-half of the upper tear attached to the tendinous portion of the subscapularis. Currently, debridement or repair is under way. But evidence-based studies are lacking and no clear treatment guidelines are available.

ELIGIBILITY:
Inclusion Criteria:

* Subscapularis tendon tear from more than 1/2 to entire of 1st facet found during routine arthroscopy with 70 degree scope
* Isolated or combined with Supraspinatus and/or Infraspinatus tear (SS/IS tear less than 3 cm)
* Combined biceps lesion
* Combined acromial clavicle (AC) arthritis

Exclusion Criteria:

* Revision case or previous surgical history of the index shoulder
* Any open surgery, including open repair of the subscapularis tendon
* Compensation case
* Combined severe arthritis of the glenohumeral joint
* Patient who selects one's own surgical method, i.e. not randomized
* Infection, tumor, etc

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2014-11-30 (Actual); Study Completion 2017-07-01 (Estimated)

PRIMARY OUTCOMES:
Range of Motion (ROM) | 2 year postoperatively
Pain Visual Analogue Scale (PVAS) | 2 year postoperatively
American Shoulder and Elbow Surgeons' score | 2 year postoperatively
Constant score | 2 year postoperatively
Korean Shoulder Score (KSS) score | 2 year postoperatively

SECONDARY OUTCOMES:
repair integrity analysis using postoperative MRI | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Burkhart SS, Tehrany AM. Arthroscopic subscapularis tendon repair: Technique and preliminary results. Arthroscopy. 2002 May-Jun;18(5):454-63. doi: 10.1053/jars.2002.30648. PMID 11987054
- [Background] Denard PJ, Jiwani AZ, Ladermann A, Burkhart SS. Long-term outcome of a consecutive series of subscapularis tendon tears repaired arthroscopically. Arthroscopy. 2012 Nov;28(11):1587-91. doi: 10.1016/j.arthro.2012.02.031. Epub 2012 May 24. PMID 22632896
- [Background] Flury MP, John M, Goldhahn J, Schwyzer HK, Simmen BR. Rupture of the subscapularis tendon (isolated or in combination with supraspinatus tear): when is a repair indicated? J Shoulder Elbow Surg. 2006 Nov-Dec;15(6):659-64. doi: 10.1016/j.jse.2005.07.013. Epub 2006 Oct 19. PMID 17055750
- [Derived] Jeong JY, Kim SC, Lee SM, Yoo JC. Prospective Randomized Clinical Trial of Arthroscopic Repair Versus Debridement for Partial Subscapularis Tendon Tears More Than Half of the Entire First Facet. Am J Sports Med. 2023 Sep;51(11):2804-2814. doi: 10.1177/03635465231187033. Epub 2023 Aug 7. PMID 37548022